CLINICAL TRIAL: NCT00541788
Title: Evaluation of the Efficacy and Safety of Common Sage in Controlling Hot Flashes in Prostate Cancer Patients Treated by Androgen Deprivation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Farmafyt (Unknown)
Responsible Party: Gert De Meerleer, MD, PhD, University Hospital Ghent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007/285
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Administration of Common Sage
  Interventions: Other: Administration of Common Sage

INTERVENTIONS:
Other: Administration of Common Sage — Administration of Common Sage

SUMMARY:
The purpose of this clinical phase I study is to measure the efficacy and side effects of Common Sage in the treatment of hot flashes in 10 patients with prostate cancer who receive androgen deprivation (AD) (exclusively or as part of a multimodality treatment) for a period of minimum 6 months. Concomitant use of a non-steroidal anti-androgen during the first month of the AD is permitted to prevent the flair-up phenomenon. However, the inclusion of patients in the study will only start at least 2 weeks after the cessation of the anti-androgen. This is done to exclude a possible influence of the anti-androgen on the severity and frequency of hot flashes.

Once the informed consent is signed, the patient receives the study diary to note the daily frequency and severity of hot flashes and their effect on daily quality of life. The severity of the hot flashes is measured by the Moyad scoring scale. The effect on daily quality of life is measured using the Hot Flash Related Daily Interference Scale (HFRDIS). The patient will be instructed in detail how to use the diary.

After week 1, the patient returns the diary to the responsible physician. In return the patient receives the study medication (Common Sage, product) and a diary for the next week (=week 2). This procedure will be repeated until the end of the observation period (2 months after enrollment in the study). The common Sage will be provided in tablets. The suggested dose of Common Sage is 3 tablets a day (morning - noon - evening).

To be sure that the effect of Common Sage is NOT due to an inhibition of the effect of the LHRH analogue, the related hormones (testosterone, FSH, LH, free testosterone and SHBG) will be tested at three fixed moments: day of study enrollment, 1 month after study enrollment and at the end of the study. In order to check the level of hemoglobin and cholesterol, every 2 weeks a blood count will be performed. It has been shown that LHRH analogues can induce anemia and hypercholesterolemia. The investigators want to measure a possible effect of Common Sage on both.

There are no known side-effects of the use of Common Sage. All symptoms that could be related to the use of Common Sage will be recorded in detail. Therefore, a clinical examination including blood pressure registration will be performed by the responsible physician on a weekly base.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients treated with androgen deprivation and experiencing hot flashes.
* Karnofsky performance status ≥70%
* Age ≥18 years
* Informed consent obtained, signed and dated before specific protocol procedures

Exclusion Criteria:

* Other therapy for hot flashes
* Mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study
* Patient unlikely to comply with protocol, i.e. uncooperative attitude, inability to complete the diary, inability to return for follow-up visits, and unlikely to complete the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Scoring of virtual side effects. | 2 months after enrollment

SECONDARY OUTCOMES:
Improvement of QOL following HFRDIS. | 2 months after enrollment
Registration of virtual side effects. | 2 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Gert De Meerleer, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be